CLINICAL TRIAL: NCT06767904
Title: A Protocol for a Randomized Trial Comparing the Efficacy of Exertional Oxygen Delivery by Continuous Versus Demand-Based Flow Systems During Six-minute Walk Test in Patients With Fibrotic Interstitial Lung Disease and Chronic Obstructive Pulmonary Disease (OXYCODE)
Brief Title: Continuous Versus Demand-Based Oxygen in Patients With Fibrotic Interstitial Lung Disease and Chronic Obstructive Pulmonary Disease
Acronym: OXYODE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sissel Kronborg-White (Other)
Responsible Party: Sponsor-Investigator, Sissel Kronborg-White, Pulmonologist, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: OXYCODE
Record Dates: First submitted 2025-01-05; First posted 2025-01-10 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Interstitial Lung Disease; Chronic Obstructive Pulmonary Disease
Keywords: Interstitial Lung Disease; Chronic Obstructive Pulmonary Disease; Oxygen Therapy; Palliation
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continous oxygen (Other): Oxygen delivery by Continous Oxygen Bottles
  Interventions: Device: Continous Oxygen by Bottles
- Demand Based Oxygen (Other): Oxygen Delivery by Demand Oxygen delivery system.
  Interventions: Device: Demand oxygen by Portable Concentrator

INTERVENTIONS:
Device: Continous Oxygen by Bottles — Oxygen delivery by bottles giving a continous flow.
  Arms: Continous oxygen
Device: Demand oxygen by Portable Concentrator — Oxygen delivery by consentrators, giving oxygen only when inhaling.
  Arms: Demand Based Oxygen

SUMMARY:
The goal of this randomised clinical trial is to compare the efficacy of exertional oxygen delivery by continous versus demand-based flow systems in patients with fibrotic Interstitial lung disease and chronic obstructive pulmonary disease . The main questions it aim to answer:

Is there a difference in lowest oxygen saturation? Is there a difference in saturation: time below <90%, pulse rate, distance and patient preferences ? It is a cross over study, so all patients will test both methods. Participants will perform 2 6-minute walk tests with the two different oxygen delivery systems.

DETAILED DESCRIPTION:
The study design is a single center, randomized, open-label cross-over exploratory comparative study to investigate the efficacy of two different oxygen delivery systems. Patients with chronic obstructive Pulmonary disease or fibrotic Interstitial Lung Disease that during a six-minute walk test can walk at least 50 m and desaturate below 88%, can be included in the study. The participants are performing 2 6-minute walk tests, randomized to perform the test with oxygen bottles or portable concentrators first. Primary endpoint is the difference in the lowest oxygen saturation between the two systems. Secondary endpoints are amongst others: difference in percentage of time and number of minutes when oxygen falls below 90%, mean and maximum pulse rate, distance and time taken to recover during the 6-minute walk test and scores from questionnaires. After 3-6 months, semistructured interviews will be done to record participants' experiences of ambulatory oxygen therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Verified diagnosis of fibrotic interstitial lung disease or chronic obstructive pulmonary disease
* Desaturation < 88% during 6-minute walk test or currently receiving ambulatory oxygen by continous oxygen
* Able to walk at least 50 meters during a 6-minute walk test
* Self-reported stable respiratory symptoms in the previous 2 weeks
* Cognitively able to understand and participate in the study
* Written informed consent

Exclusion Criteria:

* Any physical condition including paralysis, lower extremity pain, or other musculoskeletal problems limiting exercise performance
* Unstable heart condition or symptomatic stenotic valve disease
* Smoking during the previous 24 hours
* Pregnant women
* Anemia, Hb < 7.3 mmol/l (women) or < 8.3 mmol/l (men)
* Non-invasive ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Lowest oxygen | At Baseline
  difference in the lowest oxygen saturation between the two different oxygen delivery systems during a 6-min. walk test.

SECONDARY OUTCOMES:
percentage of saturation <90% | At baseline
  Percentage of time when oxygen levels fall below 90% during walk test.
minutes of saturation <90% | At baseline
  Number of minutes when saturation falls below 90% during walk test.
minimum value of oxygen | At baseline
  Minimum value of oxygen saturation during walk test
Pulse rate | At baseline
  Mean pulse rate during walk test
Maximum pulse rate | At baseline
  Maximum pulse rate during walk test
Distance | At baseline
  Difference in walk test distance
time to recover | At baseline
  The time taken to recover oxygen saturation after walk test to the level obtained at rest
Maximal Borg scale | At baseline
  Maximal rating of dyspnea on the Borg scale (Borg Rating of Percived exertion, range 0-10, where 10 is maximal breathing difficulty).
Change Borg scale | At baseline
  Change in dyspnea from rest to end of the walk test measured by the Borg scale. (Borg Rating of Percived exertion, range 0-10, where 10 is maximal breathing difficulty)
Patient preference | At baseline
  Patient preferences for the two different systems ("Which system do you prefer?"
Comfort Likert scale | At baseline
  Comfort measured by a Likert scale on a scale from 1-7 where 1 equals strongly disagree and 7 equals strongly agree. There is no unabbreviated scale title.
Reliability Likert scale | At baseline
  Reliability measured by a Likert scale on a scale from 1-7 where 1 equals strongly disagree and 7 equals strongly agree. There is no unabbreviated scale title.
Semi structured qualitative interviews | After 3-6 months
  Semi-structured qualitative interviews about patients' view on the different oxygen delivery systems
comfort and frequency use oxygen | After 3-6 months
  Questions regarding the use of the oxygen delivery systems with respect to comfort and frequency of use
Quality of life questionnaire score | After 3-6 months
  Change on Quality of life questionnaires between baseline and three to six months
Baseline Characteristics | After 3-6 months
  Associations between baseline characteristics and effect of and patient views on oxygen delivery systems

CONTACTS AND LOCATIONS:
Overall Officials: Sissel Kronborg-White, MD, PhD, Principal Investigator — Aarhus University Hospital

IPD SHARING:
Plan to Share IPD: Yes
Full access to the protocol, participants dataset and statistical codes will be granted on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Full access to the protocol, participants dataset and statistical codes will be granted on reasonable request for up to 5 years after the study has ended.
Access Criteria: Full access to the protocol, participants dataset and statistical codes will be granted on reasonable request.

REFERENCES:
- [Derived] Kronborg-White S, Jensen JH, Bendstrup E, Prior TS. Comparing the efficacy of exertional oxygen delivery by continuous versus demand-based flow systems during 6-minute walk test in patients with fibrotic interstitial lung disease and COPD in a hospital setting (OXYCODE): a protocol for a randomised trial. BMJ Open. 2025 May 16;15(5):e099664. doi: 10.1136/bmjopen-2025-099664. PMID 40379312